CLINICAL TRIAL: NCT06606353
Title: Talk-to-Jo" Intelligent Digital Health Companion, Neurocognitive Disorders and Dyads: a Qualitative Study
Brief Title: Talk-to-Jo" Intelligent Digital Health Companion, Neurocognitive Disorders and Dyads
Status: Recruiting | Type: Observational
Sponsor: Olivier Beauchet (Other Government)
Collaborators: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Sponsor-Investigator, Olivier Beauchet, MD PhD, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Organization: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Other Study IDs: 2025-2225
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Caregiver; Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dyad: people with neurocognitive disorders and their carers with an intelligent digital health companion
  Interventions: Behavioral: Talk-To-Jo

INTERVENTIONS:
Behavioral: Talk-To-Jo — Participation begins with the completion of a socio-demographic questionnaire. Next, participants test the Talk-to-Jo intelligent digital health companion on a tablet: first, a member of the research team explains the tool to the dyad (person with a neurocognitive disorder and their caregiver). The person with the disorder then interacts with Talk-to-Jo, possibly with the help of their caregiver. An observer is present, but does not intervene unless there are questions or technical problems. At the end of the test, health recommendations are given. Questions focus on the participant's memory and depression.
  Next, a 30-minute interview is conducted with a member of the research team to gather impressions of the tool, digital skills, barriers and facilitators to using AI, as well as your expectations of Talk-to-Jo.
  An additional individual interview can be arranged if required.

SUMMARY:
By 2050, one in six people in the world will be over 65, leading to an increase in the number of people with neurocognitive disorders (NCD), such as Alzheimer's disease. The number of cases will rise from 57 million to 153 million by 2050. This presents challenges for healthcare systems, as NCDs affect not only mental health but also the physical health, psychological well-being, and social relationships of patients, as well as their caregivers (PCA).

In Quebec, primary care is often inadequate for people living with NCDs due to delays in accessing resources, incomplete coverage of needs, and the COVID-19 pandemic, which has exacerbated these challenges. This situation can lead to a deterioration in patients' health, affecting their quality of life as well as that of their PCAs, while also increasing healthcare costs.

Many elderly people wish to age at home, but cognitive and functional decline complicates this desire. PCAs, generally family members or close friends, play an essential role in the daily support of these individuals. Their role, as defined in the Act to support caregivers in Quebec, includes non-professional and voluntary assistance to improve the quality of life of the person being cared for.

However, the support provided by PCAs can lead to significant stress, especially if public services are insufficient. The exhaustion of PCAs is often correlated with the severity of the care recipient's loss of autonomy. This exhaustion impacts the mental and physical health of PCAs, leading to isolation, depression, and anxiety, as well as reduced productivity and an increase in sick leave. It is therefore urgent to find support solutions to prevent PCA burnout.

Telehealth, which involves remote consultations through information and communication technologies (ICT), appears to be a promising solution to improve access to care for people with NCDs, especially in underserved areas. By enabling remote monitoring, telehealth facilitates aging in place while stimulating the remaining capacities of patients, such as responsiveness to sensory stimuli.

Artificial intelligence (AI) is also a promising tool for tracking the health of older adults in real-time, detecting early signs of diseases, and providing personalized recommendations. Virtual assistants or avatars, like "Talk-to-Jo," can interact with patients to reduce their sense of loneliness. However, the effectiveness of these technologies depends on their accessibility and adaptability to the needs of patients, particularly in cases of sensory impairments.

"Talk-to-Jo" is a digital avatar designed for older adults with NCDs and their PCAs. It asks questions about memory and depression and provides tailored recommendations to prevent or stabilize detected disorders. A first version of this tool is currently available on a tablet.

With the growing number of people living with NCDs, it is essential to develop support solutions based on telemedicine and AI. It is important to assess the usability and acceptability of these technologies by patients and their PCAs to ensure their effectiveness.

ELIGIBILITY:
1. Person living with an neurocognitive disorder (NCD):

   1. Inclusion criteria:

      * Be 65 years old or older.
      * Have an NCD, whether minor or major, in a mild to moderate stage, diagnosed within the past year.
      * Be receiving care for an NCD at the outpatient clinic of the Montreal Geriatric University Institute.
      * Have a caregiver.
      * Live in a personal residence or in a non-medicalized senior residence.
      * Be able to understand spoken and written French. The "Talk-to-Jo" avatar has only been developed in the French language and can only communicate and understand French.
   2. Exclusion criteria:

      * Inability to provide informed consent for participation in the study.
      * Participating in a concurrent experimental clinical study, to avoid interference with our study.
      * Living in a Long-Term Care Facility or in a medicalized section of an non-medicalized senior residence.
      * Inability to understand spoken and written French.
      * Having a moderate to severe visual or auditory impairment. The criterion for assessing hearing impairment will be the person's ability to understand and participate in a phone conversation. Individuals with impairments who use hearing aids or glasses to compensate for the impairments may be included.
2. Caregiver

   1. Inclusion criteria:

      * Be a caregiver for a person living with an NCD (regardless of the relationship: spouse, child, friend, neighbor, family member).
      * Be able to understand spoken and written French.
   2. Exclusion criteria:

      * Have an NCD.
      * Inability to understand spoken and written French.
      * Participating in a concurrent experimental clinical study, to avoid interference with our study.
      * Having a moderate to severe visual or auditory impairment. The criterion for assessing hearing impairment will be the person's ability to understand and participate in a phone conversation. Individuals with impairments who use hearing aids or glasses to compensate for the impairments may be included.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: dyads composed of people living with NCD and their caregiver
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
usage behaviours | Intervention day, during 15 minutes
  Semi-directed interviews will be conducted with both members of the dyad and by one or two members of the research team. If members of the research team observe a difference of opinion between the two members of the dyad, a complementary semi-structured interview will be conducted with each member of the dyad separately. This complementary semi-structured interview will take place if the members of the dyad agree to be separated for 10 to 15 minutes.
impressions and feedback from people living with an NCD and their caregivers (PPA) | Intervention day, during 15 minutes
  Semi-directed interviews will be conducted with both members of the dyad and by one or two members of the research team. If members of the research team observe a difference of opinion between the two members of the dyad, a complementary semi-structured interview will be conducted with each member of the dyad separately. This complementary semi-structured interview will take place if the members of the dyad agree to be separated for 10 to 15 minutes.
enablers and barriers to the use of the intelligent digital avatar "Talk-to-Jo." | Intervention day, during 15 minutes
  Semi-directed interviews will be conducted with both members of the dyad and by one or two members of the research team. If members of the research team observe a difference of opinion between the two members of the dyad, a complementary semi-structured interview will be conducted with each member of the dyad separately. This complementary semi-structured interview will take place if the members of the dyad agree to be separated for 10 to 15 minutes.
expectations and needs of people living with an NCD and their caregivers | Intervention day, during 15 minutes
  Semi-directed interviews will be conducted with both members of the dyad and by one or two members of the research team. If members of the research team observe a difference of opinion between the two members of the dyad, a complementary semi-structured interview will be conducted with each member of the dyad separately. This complementary semi-structured interview will take place if the members of the dyad agree to be separated for 10 to 15 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided